CLINICAL TRIAL: NCT01523171
Title: A Phase II, Multicenter, Open Label, Single Arm Study of SAR302503 in Subjects Previously Treated With Ruxolitinib and With a Current Diagnosis of Intermediate or High-Risk Primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis, or Post-Essential Thrombocythemia Myelofibrosis
Brief Title: Phase II, Open Label, Single Arm Study of SAR302503 In Myelofibrosis Patients Previously Treated With Ruxolitinib
Acronym: JAKARTA2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARD12181; 2011-005226-21 (EudraCT Number); U1111-1124-0967 (Other: UTN)
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2016-02

CONDITIONS: Hematopoietic Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAR302503 400 mg (Experimental): once daily in consecutive 28-day cycles, flexible dosing regimen (the starting dose is 400mg/day), orally, empty stomach, approximately same time each day
  Interventions: Drug: SAR302503

INTERVENTIONS:
Drug: SAR302503 — Pharmaceutical form:capsule
  Route of administration: oral

SUMMARY:
Primary Objective:

- To evaluate the efficacy of once daily dose of SAR302503 in subjects previously treated with ruxolitinib and with a current diagnosis of intermediate-1 with symptoms, Intermediate-2 or high-risk primary myelofibrosis (PMF), post-polycythemia vera myelofibrosis (Post-PV MF), or post-essential thrombocythemia myelofibrosis (Post-ET MF) based on the reduction of spleen volume at the end of 6 treatment cycles;

Secondary Objectives:

* To evaluate the effect of SAR302503 on Myelofibrosis (MF) associated symptoms as measured by the modified Myelofibrosis Symptom Assessment Form (MFSAF) diary
* To evaluate the durability of splenic response
* To evaluate the splenic response to SAR302503 by palpation at the end of Cycle 6
* To evaluate the splenic response to SAR302503 at the end of Cycle 3
* To evaluate the effect of SAR302503 on the Janus kinase 2 (JAK2) V617F allele burden
* To evaluate the safety and tolerability of SAR302503 in this population
* To evaluate plasma concentrations of SAR302503 for population PK analysis, if warranted

DETAILED DESCRIPTION:
The expected duration of the treatment in this study is approximately 8 months, based on a maximum 28-day screening period, followed by a 6-month (6-cycle) treatment period, and an EOT visit for subjects who will not continue the treatment after completing the 6 cycles of SAR302503, or discontinue the treatment early for any reasons as well as a follow-up visit which should occur 30 days after the last administration of SAR302503. Patients who continue to benefit clinically will be allowed to remain on study medication beyond the 6-month treatment period until the occurrence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of PMF or Post-PV MF or Post-ET MF, according to the 2008 World Health Organization and IWG-MRT response criteria
* Subjects who previously received Ruxolitinib treatment for PMF or Post-PV MF or Post-ET MF or PV or ET for at least 14 days (exposure of <14 days is allowed for subjects who discontinued Ruxolitinib due to intolerability or allergy) and discontinued the treatment for at least 14 days prior to the first dose of SAR302503
* MF classified as Intermediate-1 with symptoms, Intermediate-2 or high-risk by Dynamic International Prognostic Scoring System (Passamonti et al., Blood 2010)
* Spleen ≥5 cm below costal margin as measured by palpation
* Male and female subjects ≥18 years of age
* Signed written informed consent

Exclusion criteria:

* Splenectomy
* Eastern Cooperative Oncology Group (ECOG) performance status of >2 before the first dose of SAR302503 at Cycle 1 Day1
* The following laboratory values within 14 days prior to the initiation of SAR302503:

  * Absolute Neutrophil Count (ANC) <1.0 x 10exp9/L
  * Platelet count <50 x 10exp9/L
  * Serum creatinine >1.5 x Upper limit of normal (ULN)
  * Serum amylase and lipase >1.5 x ULN
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2.5 x ULN
* Total bilirubin ≥3.0 x ULN
* Subjects with total bilirubin between 1.5-3.0 x ULN must be excluded if the direct bilirubin fraction is ≥25% of the total
* Subjects with known active (acute or chronic) Hepatitis A, B, or C; and Hepatitis B and C carriers
* Prior history of chronic liver disease (eg, chronic alcoholic liver disease, autoimmune hepatitis, sclerosing cholangitis, primary biliary cirrhosis, hemachromatosis, non-alcoholic steatohepatitis [NASH])
* Subjects with any other prior malignancies are not eligible, except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which subject has been disease-free for at least 5 years
* Any chemotherapy, immunomodulatory drug therapy (eg, thalidomide, interferon-alpha), Anagrelide, immunosuppressive therapy, corticosteroids >10 mg/day prednisone or equivalent, or growth factor treatment (eg, erythropoietin), or hormones (eg, androgens, danazol) within 14 days prior to initiation of SAR302503; darbepoetin use within 28 days prior to initiation of SAR302503.The only chemotherapy allowed will be hydroxyurea within 1 day prior to initiation of SAR302503
* Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of SAR302503

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Response Rate (RR), defined as the proportion of subjects who have a ≥35% reduction from baseline in volume of spleen at the end of Cycle 6 as measured by Magnetic Resonance Imaging (MRI) (or CT scan in subjects with contraindications for MRI) | 6 months

SECONDARY OUTCOMES:
Symptom Response Rate (SRR): Proportion of subjects with a ≥50% reduction from baseline to the end of Cycle 6 in the total symptom score using the modified MFSAF | 6 months
Duration of spleen response, measured by MRI (or CT scan in subjects with contraindications for MRI) | 6 months
Proportion of subjects with a ≥50% reduction in length of spleen by palpation from baseline at the end of Cycle 6 | 6 months
Response Rate at the end of Cycle 3, defined as the proportion of subjects who have a ≥35% reduction from baseline in volume of spleen at the end of Cycle 3 as measured by MRI (or CT scan in subjects with contraindications for MRI) | 6 months
Percent change of spleen volume at the end of Cycles 3 and 6 from baseline as measured by MRI (or CT scan in subjects with contraindications for MRI) | 6 months
Safety, as assessed by clinical, laboratory, ECG, and vital sign events; graded by the NCI CTCAE v4.03 | approximately 5 years
Plasma concentrations of SAR302503 | 4 months
The effect of SAR302503 on the JAK2V617F allele burden | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (42):
- United States (16):
  - Investigational Site Number 840007, Phoenix, Arizona
  - Investigational Site Number 840003, San Francisco, California
  - Investigational Site Number 840004, San Francisco, California
  - Investigational Site Number 840005, Atlanta, Georgia
  - Investigational Site Number 840014, Chicago, Illinois
  - Investigational Site Number 840001, Kansas City, Kansas
  - Investigational Site Number 840017, Baltimore, Maryland
  - Investigational Site Number 840013, Baltimore, Maryland
  - Investigational Site Number 840010, Ann Arbor, Michigan
  - Investigational Site Number 840009, New York, New York
  - Investigational Site Number 840018, New York, New York
  - Investigational Site Number 840022, Cleveland, Ohio
  - Investigational Site Number 840019, Middletown, Ohio
  - Investigational Site Number 840024, Charleston, South Carolina
  - Investigational Site Number 840002, Houston, Texas
  - Investigational Site Number 840015, Salt Lake City, Utah
- Austria (2):
  - Investigational Site Number 040002, Salzburg
  - Investigational Site Number 040001, Vienna
- Belgium (2):
  - Investigational Site Number 056002, Antwerp
  - Investigational Site Number 056003, Leuven
- Investigational Site Number 124001, Toronto, Canada
- France (5):
  - Investigational Site Number 250001, Marseille
  - Investigational Site Number 250003, Nîmes
  - Investigational Site Number 250002, Paris
  - Investigational Site Number 250006, Paris
  - Investigational Site Number 250004, Toulouse
- Germany (5):
  - Investigational Site Number 276003, Frankfurt am Main
  - Investigational Site Number 276007, Leipzig
  - Investigational Site Number 276006, Magdeburg
  - Investigational Site Number 276001, Mannheim
  - Investigational Site Number 276005, Ulm
- Italy (4):
  - Investigational Site Number 380004, Florence
  - Investigational Site Number 380001, Milan
  - Investigational Site Number 380002, Roma
  - Investigational Site Number 380003, Varese
- Netherlands (3):
  - Investigational Site Number 528002, Amsterdam
  - Investigational Site Number 528003, Maastricht
  - Investigational Site Number 528001, Nijmegen
- Spain (3):
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724003, Majadahonda
  - Investigational Site Number 724002, Salamanca
- Investigational Site Number 826001, London, United Kingdom

REFERENCES:
- [Derived] Harrison CN, Schaap N, Vannucchi AM, Kiladjian JJ, Tiu RV, Zachee P, Jourdan E, Winton E, Silver RT, Schouten HC, Passamonti F, Zweegman S, Talpaz M, Lager J, Shun Z, Mesa RA. Janus kinase-2 inhibitor fedratinib in patients with myelofibrosis previously treated with ruxolitinib (JAKARTA-2): a single-arm, open-label, non-randomised, phase 2, multicentre study. Lancet Haematol. 2017 Jul;4(7):e317-e324. doi: 10.1016/S2352-3026(17)30088-1. Epub 2017 Jun 8. PMID 28602585